CLINICAL TRIAL: NCT05048589
Title: Feasibility of Randomizing Danish Citizens Aged 65-79 Years to High-Dose Quadrivalent Influenza Vaccine vs. Standard-Dose Quadrivalent Influenza Vaccine in a Pragmatic Registry-Based Setting
Acronym: DANFLU-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tor Biering-Sørensen (Other)
Collaborators: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor-Investigator, Tor Biering-Sørensen, Research Director, MD, PhD, MPH, Herlev and Gentofte Hospital
Organization: Herlev and Gentofte Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DANFLU-1; QHD00027 (Other: Sanofi Pasteur); 2021-003170-31 (EudraCT Number)
Record Dates: First submitted 2021-08-31; First posted 2021-09-17 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Influenza
Keywords: Influenza; Vaccination; Pragmatic; Registry
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard-Dose Quadrivalent Influenza Vaccine (Active Comparator): QIV-SD single injection at Day 0
  Interventions: Drug: Standard-Dose Quadrivalent Influenza Vaccine
- High-Dose Quadrivalent Influenza Vaccine (Experimental): QIV-HD single injection at Day 0
  Interventions: Drug: High-Dose Quadrivalent Influenza Vaccine

INTERVENTIONS:
Drug: Standard-Dose Quadrivalent Influenza Vaccine — For the control arm, the standard-dose quadrivalent influenza vaccines Influvactetra® and Vaxigriptetra will be used.
  Other Names: QIV-SD
  Arms: Standard-Dose Quadrivalent Influenza Vaccine
Drug: High-Dose Quadrivalent Influenza Vaccine — For the control arm, the high-dose quadrivalent influenza vaccine Efluelda®/Fluzone® High-Dose Quadrivalent will be used.
  Other Names: QIV-HD
  Arms: High-Dose Quadrivalent Influenza Vaccine

SUMMARY:
The purpose of the study is to assess the feasibility of identifying, recruiting and randomizing a large sample of Danish citizens aged 65-79 years to high-dose quadrivalent influenza vaccine or standard-dose quadrivalent influenza vaccine in the 2021/2022 influenza season in a registry-based setting using Danish nationwide registries for all data collection including baseline information and outcome assessment.

DETAILED DESCRIPTION:
To evaluate the feasibility of recruiting and randomizing Danish citizens aged 65-79 years, we aim to randomize 40,000 citizens 1:1 to high-dose quadrivalent influenza vaccine or standard-dose quadrivalent influenza vaccine in a pragmatic, open-label, registry-based design using the infrastructure of Danske Lægers Vaccinations Service (DLVS), an organization responsible for numerous vaccination clinics in Denmark, for recruitment and randomization and Danish nationwide registries for data collection. Citizens will be recruited by DLVS and randomized and vaccinated at the DLVS clinics. All collection of data related to baseline information, outcomes, and safety monitoring will be performed by a central trial site utilizing information from Danish nationwide health registries.

The findings of this pilot trial will indicate whether the conduction of a full-scale, adequately powered pragmatic RCT is feasible within the Danish registry-based framework.

ELIGIBILITY:
Inclusion Criteria:

1. Age 65-79 years
2. Informed consent form has been signed and dated

Exclusion Criteria:

1. Allergy/hypersensitivity towards the influenza vaccines used in this study

Ages: 65 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 12551 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Number of persons contacted by recruitment letter | Up to 8 months
Number of participants included and randomized to QIV-HD or QIV-SD | Up to 8 months
Agreement between randomization assignment and actual received vaccine | Up to 8 months
Balance between groups in terms of number of subjects in each arm and baseline characteristics | Up to 8 months
Comparison of baseline characteristics for the QIV-HD and QIV-SD groups to the overall Danish general population aged 65-79 years | Up to 8 months
Comparison of baseline characteristics for the QIV-HD and QIV-SD groups to the population aged 65-79 years in the DLVS database used for recruitment | Up to 8 months
Description of event rates and calculation of relative vaccine effectiveness for hospitalization for influenza and/or pneumonia | >= 14 days after vaccination up to 8 months post-vaccination
  First hospitalization with a primary (A) diagnosis code for influenza or pneumonia of at least 1 night duration
Description of event rates and calculation of relative vaccine effectiveness for hospitalization for respiratory disease | >= 14 days after vaccination up to 8 months post-vaccination
  First hospitalization with a primary (A) diagnosis code for respiratory disease of at least 1 night duration
Description of event rates and calculation of relative vaccine effectiveness for hospitalization for cardio-respiratory disease | >= 14 days after vaccination up to 8 months post-vaccination
  First hospitalization with a primary (A) diagnosis code for cardio-respiratory disease of at least 1 night duration
Description of event rates and calculation of relative vaccine effectiveness for hospitalization for cardiovascular disease | >= 14 days after vaccination up to 8 months post-vaccination
  First hospitalization with a primary (A) diagnosis code for cardiovascular disease of at least 1 night duration
Description of event rates and calculation of relative vaccine effectiveness for hospitalization from any cause | >= 14 days after vaccination up to 8 months post-vaccination
  First hospitalization with any diagnosis code of at least 1 night duration
Description of event rates and calculation of relative vaccine effectiveness for all-cause mortality | >= 14 days after vaccination up to 8 months post-vaccination
  Death from any cause
Description of event rates and calculation of relative vaccine effectiveness for hospitalization for COVID-19 | >= 14 days after vaccination up to 8 months post-vaccination
  First hospitalization with a primary (A) diagnosis code for COVID-19 of at least 1 night duration

CONTACTS AND LOCATIONS:
Overall Officials: Tor Biering-Sørensen, MD, PhD, MPH, Study Chair — Research Director
Locations (2):
- Denmark (2):
  - Cardiovascular Non-Invasive Imaging Research Laboratory, Department of Cardiology, Herlev and Gentofte Hospital, Hellerup
  - Danske Lægers Vaccinations Service, Søborg

IPD SHARING:
Plan to Share IPD: No
Sharing of individual-level data stemming from Danish administrative registries is illegal according to Danish law.

REFERENCES:
- [Derived] Langhoff AF, Johansen ND, Modin D, Janstrup KH, Bartholdy KV, Espersen C, Nealon J, Samson S, Loiacono MM, Harris R, Larsen CS, Jensen AMR, Landler NE, Claggett BL, Solomon SD, Landray MJ, Gislason GH, Kober L, Sivapalan P, Jensen JUS, Biering-Sorensen T. High-Dose vs. Standard-Dose Influenza Vaccine in Older Patients With Hypertension: A Post Hoc Analysis of DANFLU-1. J Clin Hypertens (Greenwich). 2025 Nov;27(11):e70177. doi: 10.1111/jch.70177. PMID 41238377
- [Derived] Duus LS, Johansen ND, Modin D, Janstrup KH, Nealon J, Samson S, Loiacono MM, Harris RC, Larsen CS, Reimer Jensen AM, Claggett BL, Solomon SD, Landray MJ, Gislason GH, Kober L, Sivapalan P, Staehr Jensen JU, Biering-Sorensen T. Effects of high-dose versus standard-dose influenza vaccine among patients with chronic lung disease: A prespecified analysis of the DANFLU-1 trial. Respir Investig. 2025 Nov;63(6):1309-1315. doi: 10.1016/j.resinv.2025.10.016. Epub 2025 Nov 1. PMID 41177098
- [Derived] Christensen J, Johansen ND, Janstrup KH, Modin D, Skaarup KG, Nealon J, Samson S, Loiacono M, Harris R, Larsen CS, Jensen AMR, Landler NE, Claggett BL, Solomon SD, Gislason GH, Kober L, Landray MJ, Sivapalan P, Jensen JUS, Biering-Sorensen T. Time of day for vaccination, outcomes, and relative effectiveness of high-dose vs. standard-dose quadrivalent influenza vaccine: A post hoc analysis of the DANFLU-1 randomized clinical trial. J Infect. 2024 Nov;89(5):106276. doi: 10.1016/j.jinf.2024.106276. Epub 2024 Sep 18. PMID 39303788
- [Derived] Christensen J, Johansen ND, Modin D, Janstrup KH, Nealon J, Samson S, Loiacono M, Harris R, Larsen CS, Jensen AMR, Landler NE, Claggett BL, Solomon SD, Gislason GH, Kober L, Landray MJ, Sivapalan P, Jensen JUS, Biering-Sorensen T. Relative Effectiveness of High-Dose Versus Standard-Dose Quadrivalent Influenza Vaccine in Older Adults With Cardiovascular Disease: A Prespecified Analysis of the DANFLU-1 Randomized Clinical Trial. Circ Cardiovasc Qual Outcomes. 2025 Feb;18(2):e011496. doi: 10.1161/CIRCOUTCOMES.124.011496. Epub 2024 Aug 31. PMID 39215646
- [Derived] Johansen ND, Modin D, Nealon J, Samson S, Salamand C, Loiacono MM, Larsen CS, Jensen AMR, Landler NE, Claggett BL, Solomon SD, Landray MJ, Gislason GH, Kober L, Jensen JUS, Sivapalan P, Vestergaard LS, Valentiner-Branth P, Krause TG, Biering-Sorensen T. A Pragmatic Randomized Feasibility Trial of Influenza Vaccines. NEJM Evid. 2023 Feb;2(2):EVIDoa2200206. doi: 10.1056/EVIDoa2200206. Epub 2023 Jan 23. PMID 38320035
- [Derived] Johansen ND, Modin D, Skaarup KG, Nealon J, Samson S, Dufournet M, Loiacono MM, Harris RC, Larsen CS, Jensen AMR, Landler NE, Claggett BL, Solomon SD, Landray MJ, Gislason GH, Kober L, Jensen JUS, Sivapalan P, Vestergaard LS, Valentiner-Branth P, Krause TG, Biering-Sorensen T. Effectiveness of high-dose versus standard-dose quadrivalent influenza vaccine against recurrent hospitalizations and mortality in relation to influenza circulation: A post-hoc analysis of the DANFLU-1 randomized clinical trial. Clin Microbiol Infect. 2024 Nov;30(11):1453-1459. doi: 10.1016/j.cmi.2024.01.017. Epub 2024 Jan 28. PMID 38286177
- [Derived] Johansen ND, Modin D, Nealon J, Samson S, Salamand C, Larsen CS, Claggett BL, Solomon SD, Landray MJ, Gislason GH, Kober L, Jensen JUS, Sivapalan P, Vestergaard LS, Valentiner-Branth P, Krause TG, Biering-Sorensen T. Feasibility of randomizing Danish citizens aged 65-79 years to high-dose quadrivalent influenza vaccine vs. standard-dose quadrivalent influenza vaccine in a pragmatic registry-based setting: rationale and design of the DANFLU-1 Trial. Pilot Feasibility Stud. 2022 Apr 21;8(1):87. doi: 10.1186/s40814-022-01044-w. PMID 35449028